CLINICAL TRIAL: NCT01364584
Title: Impact of Exenatide on Cardiovascular Exercise Performance in Type 2 Diabetes
Acronym: Exenatide
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Amylin Pharmaceuticals, LLC. (Industry); Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 10-0438
Record Dates: First submitted 2011-05-24; First posted 2011-06-02 (Estimated); Results first posted 2018-07-09 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Exenatide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exenatide (Experimental): Pre-dosed inject-able pen (an automatic device which injects under the skin) 10 mcg twice a day of exenatide for 2.5 months
  Interventions: Drug: Exenatide
- Placebo (Placebo Comparator): Pre-dosed inject-able pen (an automatic device which injects under the skin) 10 mcg twice a day of placebo for 2.5 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Exenatide — Subcutaneous injection 2.5 micrograms (mcg) to 10 mcg twice per day (BID)
  Other Names: Byetta
  Arms: Exenatide
Drug: Placebo — Subcutaneous injection 2.5 mcg-10 mcg BID
  Arms: Placebo

SUMMARY:
Previous research in our lab and others has established that type 2 diabetes (T2D) is associated with significantly impaired functional exercise capacity, a factor which is potentially associated with an increased risk of cardiovascular disease in those with type 2 diabetes. Of great concern, the majority of people with type 2 diabetes are sedentary and one possible reason may be that exercise, even at low levels, is perceived as being a harder effort than for nondiabetic people. Thus, treatments that may motivate patients with type 2 diabetes to be more physically active have great potential benefit.

Recent observational studies suggest that glucagon-like peptide-1 agents, such as exenatide, may have a beneficial effect on endothelial and cardiac function. Because these two factors have been shown to be associated with exercise dysfunction in type 2 diabetes, the investigators hypothesize that exenatide may improve exercise capacity in those with type 2 diabetes. The aims of this study are to (1) assess whether exenatide will improve functional exercise capacity in persons with type 2 diabetes and (2) investigate the effect of exenatide on specific metabolic, endothelial, cardiac and peripheral circulatory measures of function related to changes in exercise capacity. The Investigators primary hypothesis is that exenatide will improve functional exercise capacity in people with type 2 diabetes. Having a drug that improves exercise capacity could motivate patients to exercise more and hence be a significant benefit.

DETAILED DESCRIPTION:
Subjects will come for a total of seven testing visits, including two screening visits, during which evaluations will take place. Visits are structured as follows:

Visits 1, 2 and 3 will be completed over a four-week period.

1. After subjects review the study and give consent for study participation, a history and physical exam will be performed. In addition, the Low-level Physical Activity Recall (LoPAR) questionnaire, pulmonary function testing, and vital signs will be performed.
2. Subjects will be asked to fast prior to visit 2. Blood and urine samples will be collected for measurement of glycosylated hemoglobin(HbA1C), fasting glucose, fasting insulin, free fatty acids and microalbuminuria (these measures will be covariates in the analyses). A dietary survey will be administered for food preferences for the three day study diet administered prior to visits 3, 4, 6 and 7. Dual Energy X-ray Absorptiometry (DXA) and body composition tests will be done to ensure that groups are weight similar (using fat-free mass). Autonomic nervous system testing, a resting electrocardiogram (EKG) and familiarization bicycle test will be performed.
3. Subjects will receive a three day study diet prior to visit 3. A resting and exercise EKG will be performed on the day of the visit. Patients will have measures made of cardiac function and endothelial function on visit 3 as well using plethysmography and cardiac echo. The peak aerobic capacity (VO2max) test will be performed. Vital signs will be taken at rest.
4. Randomization: Subjects will receive a three day study diet prior to visit 4. During visit four, arterial stiffness/endothelial function will be non-invasively measured by the Sphygmocor system. Subjects will have three constant-load tests to measure oxygen (VO2) kinetics where oxygen saturation (StO2) will be measured during exercise. A resting and exercise EKG and vital signs will be performed during the visit. Subjects will be randomized to either taking exenatide or placebo and all must have been taking metformin (1-2 grams /d) for at least 3 months. Exenatide will be titrated starting at 5 mcg twice per day for two weeks then moving to 10 mcg twice per day as tolerated and the placebo dose will match this titration. During the treatment phase subjects will be given a log to keep track of their blood glucose each day. Study coordinators will contact each subject weekly to obtain these values which will be checked by the study doctors and shared with the subject's primary care physician if adjustments in other medications need to be made.
5. Week 4: Visit 5 will consist of a physical exam with a clinician as well as a blood draw and check of vital signs during exenatide treatment.
6. Week 12: After 3 months of exenatide or placebo administration, the procedures of Visit 3 will be repeated as Visit 6. Additional testing to be performed during visit 6 include a physical exam performed by a study physician, DXA scan and body composition tests to monitor any changes in body composition (fat-free mass), blood work for lab tests listed in Visit 2 and the LoPAR questionnaire.
7. Week 13: During visit 7, the testing performed during visit 4 will be repeated after 3 months of exenatide or placebo administration.

Subjects will continue exenatide or placebo treatment while completing exit testing during Weeks 12 and 13.

ELIGIBILITY:
Inclusion Criteria

* Men and women between the ages of 45 and 70 years of age
* Diagnosed with uncomplicated type 2 diabetes
* Sedentary persons (exercising not more than one time per week)
* Females who are post-menopausal
* BMI must be less than 35
* Subjects must be taking metformin for diabetes control and may also be on sulfonylurea drugs or meglitinides
* Glycosylated hemoglobin (HbA1C) <9%
* Non-smokers or former smokers who have quit for at least 1 year
* Absence of comorbid conditions
* Resting systolic blood pressure < 190, Resting diastolic blood pressure < 95

Exclusion Criteria

* People with type 2 diabetes (T2D) taking oral medications, other than metformin or sulfonylurea drugs or meglitinides, to control their diabetes.
* Persons treated with insulin will be excluded
* People who are currently smoking or have not quit for at least one year
* Peripheral neuropathy
* Regional wall motion abnormalities
* Left ventricular systolic dysfunction
* Ischemic heart disease (abnormal resting or exercise electrocardiogram)
* Presence of angina that would limit exercise performance
* Pulmonary problems that would limit exercise performance
* Systolic blood pressure >190 mmHg at rest or >250 mmHg with exercise or diastolic pressure >95 mmHg at rest or >115 mmHg with exercise
* Persons with autonomic dysfunction (>20 mm fall in upright BP without a change in heart rate)
* Proteinuria (urine protein >200 mg/dl) or a creatinine > 2.0 mg/dl
* Renal disease
* Persons with peripheral arterial disease
* Persons with a history of pancreatitis

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2010-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith G Regensteiner, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Exenatide: Pre-dosed injectable pen (an automatic device which injects under the skin) 10 mcg twice a day of exenatide for 2.5 months
  Exenatide: Subcutaneous injection 2.5 micrograms (mcg) to 10 mcg twice per day (BID)
- Placebo: Pre-dosed injectable pen (an automatic device which injects under the skin) 10 mcg twice a day of placebo for 2.5 months
  Placebo: Subcutaneous injection 2.5 mcg-10 mcg BID
Period: Overall Study
Arm/Group | Exenatide | Placebo
Started | 11 | 12
Completed | 11 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exenatide | Placebo | Total
Number analyzed (Participants) | 11 | 12 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (7) | 64 (1) | 64 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 11
  Male | 7 | 5 | 12
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11 | 12 | 23
Body Mass (kg) [Mean (Standard Deviation); unit: kilograms] | 101.7 (5.3) | 87.9 (3.3) | 93.4 (16.1)
Body Mass Index (kg/m2) [Mean (Standard Deviation); unit: kilograms per meter squared] | 33.9 (1.0) | 31.3 (1.2) | 32.3 (3.9)
Body Fat (%) [Mean (Standard Deviation); unit: percentage] | 37.7 (2.3) | 35.7 (2.2) | 36.7 (7.15)
Lean Mass (kg) [Mean (Standard Deviation); unit: kilograms] | 61.9 (3.9) | 55.8 (2.8) | 58.1 (11.6)
Fasting Glucose (mg/dl) [Mean (Standard Deviation); unit: milligrams per deciliter] | 170.5 (24.2) | 127.9 (8.0) | 147.6 (59.9)
Fasting Insulin (μU/ml) [Mean (Standard Deviation); unit: microunits per milliliter] | 29.0 (3.7) | 34.6 (6.4) | 31.0 (15.1)
HbA1c (%) [Mean (Standard Deviation); unit: percentage of glycated hemoglobin] | 7.3 (1.1) | 7.2 (0.4) | 7.2 (1.1)
Total Cholesterol (mg/dl) [Mean (Standard Deviation); unit: milligrams per deciliter] | 156.3 (9.8) | 175.3 (11.7) | 165.2 (34.9)
LDL Cholesterol (mg/dl) [Mean (Standard Deviation); unit: milligrams per deciliter] | 93.8 (6.2) | 97.6 (7.4) | 94.4 (22.1)
Triglycerides (mg/dl) [Mean (Standard Deviation); unit: milligrams per deciliter] | 156.8 (18.3) | 217.8 (58.0) | 190.1 (136.9)
Glycerol (mg/dl) [Mean (Standard Deviation); unit: milligrams per deciliter] | 1.21 (0.5) | 1.14 (0.5) | 1.16 (0.5)
Free Fatty Acids (mmol/L) [Mean (Standard Deviation); unit: millimoles per liter] | 580.8 (76.3) | 500.5 (67.8) | 546.3 (228.2)
VO2peak (ml/kg/min) [Mean (Standard Deviation); unit: milliliters per kilogram per minute] | 17.5 (1.0) | 15.4 (0.9) | 16.4 (3.1)
VO2peak (ml/min) [Mean (Standard Deviation); unit: milliliters per minute] | 1783 (129) | 1363 (95) | 1554 (415)
VO2 kinetics tau (sec) [Mean (Standard Deviation); unit: seconds] | 78.2 (6.8) | 63.3 (5.9) | 71.9 (19.1)
Circumferential Strain [Mean (Standard Deviation); unit: percentage difference in circumferences] — Measured via echocardiography, circumferential strain is calculated as the change in circumference of both the endocardium and the epicardium as compared to the relaxed circumference of those regions.
  percentage difference in circumferences | -23.7 (5.5) | -23.5 (5.0) | -23.6 (5.3)
Longitudinal Strain [Mean (Standard Deviation); unit: percentage difference in lengths] — Measured via echocardiography, longitudinal strain is calculated as the change in length of both the endocardium and the epicardium as compared to the relaxed length of those regions.
  percentage difference in lengths | -17.1 (3.9) | -19.3 (2.3) | -18.2 (3.4)
Stroke Volume (ml/beat) [Mean (Standard Deviation); unit: milliliters per beat] | 79.2 (22.7) | 82.5 (23.1) | 81.5 (23.1)

OUTCOME MEASURES:

1. Primary Outcome: Peak Oxygen Consumption (VO2 Peak)
Description: Subjects' peak oxygen consumption (VO2 peak) will be tested on a stationary bike before and after 3 months of study medication or placebo.
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: milliliters per kilogram per minute
Arm/Group | Exenatide | Placebo
Number analyzed (Participants) | 11 | 12
milliliters per kilogram per minute | 16.6 (1.1) | 16.1 (1.1)

2. Secondary Outcome: Oxygen Uptake Kinetics Steady State Tau
Description: Time to steady state oxygen consumption will be assessed in subject before and after 3 months of study medication or placebo.
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Exenatide | Placebo
Number analyzed (Participants) | 11 | 12
seconds | 71.4 (8.5) | 67.2 (2.7)

3. Secondary Outcome: Change From Baseline in Arterial Stiffness
Description: Pulse wave velocity will be measured via sphygmocor before and after 3 months of study medication or placebo.
Time Frame: Baseline and 3 months
Population: Data unable to be collected on all participants, hence the difference between the overall number of participants analyzed here and the actual number of participants who completed the study
Measure: Mean (Standard Deviation); unit: meters/second
Arm/Group | Exenatide | Placebo
Number analyzed (Participants) | 6 | 7
meters/second | -1.23 (1.27) | 0.37 (0.89)

4. Secondary Outcome: Change From Baseline in Peak Dilation of Brachial Artery Diameter
Description: Change in the response of the brachial artery to hyperemia will be assessed before and after 3 months of study medication or placebo.
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Exenatide | Placebo
Number analyzed (Participants) | 11 | 12
millimeters
  Pre-Intervention (Baseline) | 0.193 (0.045) | 0.192 (0.046)
  Post-Intervention (3 months) | 0.226 (0.057) | 0.151 (0.026)

5. Secondary Outcome: Change in (Non-invasively Measured) Deoxygenated Hemoglobin Concentration in the Vastus Lateralis During Exercise
Description: Deoxygenated hemoglobin concentration will be measured using near-infrared spectroscopy during sub-maximal exercise before and after 3 months of study drug administration.
Time Frame: Baseline and 3 months
Population: Data not collected
Arm/Group | Exenatide | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Echocardiographic Measures - Circumferential Strain
Description: Potential change in cardiac function will be assessed by echocardiography before and after 3 months of study medication or placebo.
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: % difference in circumferences
Arm/Group | Exenatide | Placebo
Number analyzed (Participants) | 11 | 12
% difference in circumferences | -25.6 (1.78) | -22.6 (1.4)

7. Secondary Outcome: Echocardiographic Measures - Longitudinal Strain
Description: as for outcome 6
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: % difference in lengths
Arm/Group | Exenatide | Placebo
Number analyzed (Participants) | 11 | 12
% difference in lengths | -18.5 (1.2) | -18.3 (0.8)

8. Secondary Outcome: Echocardiographic Measures - Stroke Volume
Description: as for outcome 6
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: mL/beat
Arm/Group | Exenatide | Placebo
Number analyzed (Participants) | 11 | 12
mL/beat | 93.3 (2.8) | 80.7 (1.9)

9. Secondary Outcome: Echocardiographic Measures - Mitral Valve E Wave Velocity
Description: as for outcome 6
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: centimeters/second
Arm/Group | Exenatide | Placebo
Number analyzed (Participants) | 11 | 12
centimeters/second | 0.61 (0.06) | 0.78 (0.06)

10. Secondary Outcome: Echocardiographic Measures - Mitral Valve E:A Wave Velocity
Description: as for outcome 6
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: centimeters/second
Arm/Group | Exenatide | Placebo
Number analyzed (Participants) | 11 | 12
centimeters/second | 0.85 (0.09) | 0.82 (0.06)

11. Secondary Outcome: Echocardiographic Measures - Mitral Valve Deceleration Time
Description: as for outcome 6
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Exenatide | Placebo
Number analyzed (Participants) | 11 | 12
milliseconds | 234.6 (17.0) | 239.8 (14.6)

12. Secondary Outcome: Echocardiographic Measures - Septal E'
Description: as for outcome 6
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: centimeters/second
Arm/Group | Exenatide | Placebo
Number analyzed (Participants) | 11 | 12
centimeters/second | 0.08 (0.01) | 0.07 (0.01)

13. Secondary Outcome: Echocardiographic Measures - Septal E:E'
Description: as for outcome 6
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Exenatide | Placebo
Number analyzed (Participants) | 11 | 12
ratio | 8.3 (0.9) | 12.6 (1.4)

14. Secondary Outcome: Echocardiographic Measures - Lateral E'
Description: as for outcome 6
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: centimeters/second
Arm/Group | Exenatide | Placebo
Number analyzed (Participants) | 11 | 12
centimeters/second | 0.09 (0.01) | 0.09 (0.01)

15. Secondary Outcome: Echocardiographic Measures - Lateral E:E'
Description: as for outcome 6
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Exenatide | Placebo
Number analyzed (Participants) | 11 | 12
ratio | 6.7 (0.6) | 8.4 (1.2)

ADVERSE EVENTS:
Arm/Group | Exenatide | Placebo
Serious Adverse Events (participants affected / at risk) | 3/11 | 0/12
Other Adverse Events (participants affected / at risk) | 0/11 | 0/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Exenatide (N=11) | Placebo (N=12)
Renal Neoplasm (Tumor on base of kidney) (Renal and urinary disorders) | 1 | 0 — A 60-year-old Caucasian male patient was diagnosed with a tumor on the base of the kidney while enrolled in the study. No action was taken regarding the blinded study therapy due to the event.
Eosinophil count increased (Blood and lymphatic system disorders) | 1 | 0 — A white male patient was hospitalized for eosinophil count increased (grade 1) while enrolled in the study. The patient initiated blinded study therapy on 04.23.13. Study therapy was discontinued due to the event, with last dose received on 10.22.13.
Bladder Papilloma (Renal and urinary disorders) | 1 | 0 — A 64-year-old white female patient was diagnosed with urothelial papilloma while enrolled in the study. Study therapy was held due to the event. The event was classified as a benign neoplasm with the bladder as the site of primary malignancy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No